CLINICAL TRIAL: NCT06017206
Title: Intraopertive Hypotension and Postoperative Cardiovascular Complications Among Chinese Elderly Patients Undergoing Oncardiac Surgery : a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Hao Li (Other)
Responsible Party: Sponsor-Investigator, Hao Li, associate chief physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: ChinaPLAGH301IOH
Record Dates: First submitted 2023-06-28; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
To explore the relationship of intraoperative hypotension and perioperative cardiovascular complications in elderly noncardiac surgical patients

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years
* Undergoing general anesthesia
* Inpatients who had noncardiac surgery between January 1, 2012 and August 31, 2019

Exclusion Criteria:

* ASA grade V
* Low-risk surgery (hysteroscopic and body surface surgery)
* Length of surgery ≤30 min
* Short operation interval (less than 3 days between procedures)
* Without intraoperative blood pressure value at 30s intervals
* Missing data on patient characteristics.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: age ≥65 years old patients
Sampling Method: Non-Probability Sample
Enrollment: 35262 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
postoperative cardiovascular complications | 2012-1~2019-8